CLINICAL TRIAL: NCT05141708
Title: Treatment Patterns and Clinical Outcomes Among Talazoparib-Treated Adults With HER2-Negative Metastatic Breast Cancer and Germline BRCA1/2 Mutations: An Observational Study Using Flatiron Electronic Health Record (EHR) Database
Brief Title: Treatment Patterns and Clinical Outcomes Among Talazoparib-Treated Adults With HER2-Negative mBC With gBRCA1/2m
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441055
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Breast Cancer; Breast Neoplasms
Keywords: Metastatic Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Talazoparib-treated adults with HER2- gBRCAm mBC: Adult patients with HER2-negative metastatic breast cancer with germline BRCA1/2 mutations who initiated talazoparib treatment in first-line or later line of therapy between January 1, 2018 and September 30, 2020.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Receipt of talazoparib as treatment for HER2-negative metastatic breast cancer with germline BRCA1/2 mutations anytime between January 1, 2018 and September 30, 2020
  Other Names: Talzenna

SUMMARY:
This non-interventional retrospective study will describe real-world treatment patterns and clinical outcomes among adults with HER2-negative metastatic breast cancer with germline BRCA1/2 mutations who initiated talazoparib as a first or later line of therapy. Patients will be identified from the Flatiron Electronic Health Record database.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Diagnosed with breast cancer (ICD-9 174.x or 175.x or ICD-10 C50x)
* At least two visits in the Flatiron database on or after January 1, 2011
* Pathology consistent with breast cancer
* Has evidence of stage IV or recurrent metastatic breast cancer with a metastatic diagnosis date on or after January 1, 2011. This includes patients who were diagnosed with stage IV at diagnosis or were diagnosed with earlier stage disease, then developed a distant metastasis later on, or had recurrence of the disease via a distant metastasis
* Confirmed receipt of talazoparib as treatment for mBC via abstraction initiated between January 1, 2018 and September 30, 2020
* HER2 negative test result on or before the start of patient's first talazoparib-containing line of therapy, as defined by Flatiron's line of therapy rules
* BRCA1, BRCA2, BRCA1 and BRCA2 germline mutation, or BRCA germline mutation not otherwise specified, identified on or before the start date of patient's first talazoparib-containing line of therapy, as defined by Flatiron's line of therapy business rules
* Age 18 years or older at the time of first talazoparib-containing line of therapy

Exclusion Criteria:

* Lacking relevant unstructured documents in the Flatiron database for review by the abstraction team
* Receipt of drug as part of a clinical trial (captured in the database as "clinical study drug" without additional information about active ingredient or whether the patient received placebo), defined as any non-cancelled order, administration, or oral episode for a drug used in a clinical trial, on or prior to start of first talazoparib line of therapy, as defined by Flatiron's line of therapy business rules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HER2-negative metastatic breast cancer with germline BRCA1/2 mutations who initiated talazoparib treatment in first-line or later line of therapy between January 1, 2018 and September 30, 2020 identified from Flatiron Health Analytic Database.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with human epidermal growth factor receptor 2 (HER2)-negative metastatic breast cancer (mBC) germline breast cancer susceptibility gene 1 or gene 2 mutations (gBRCA 1/2m), who initiated treatment with talazoparib on or after 01-Jan-2018 till 30-Sep-2020 (approximately 2.9 years) and were greater than or equal to (>=) 18 years of age during treatment initiation were observed retrospectively in this study.
Pre-assignment Details: Data from eligible participants were retrieved and observed in this retrospective chart review study from 17-December-2021 to 30-Jun-2022 (approximately 6.14 months of this study). Data of participants were retrieved from Flatiron Health Analytic Database.
Groups:
- Talazoparib: Eligible participants who initiated treatment with talazoparib as a first or later line of therapy under real-world routine clinical practice for HER2- mBC gBRCA 1/2m on or after 01-Jan-2018 were included.
Period: Overall Study
Arm/Group | Talazoparib
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included adult participants with HER2-negative mBC with gBRCA1/2 mutations who initiated talazoparib treatment in first-line or later identified from Flatiron Health Analytic Database.
Groups:
- Talazoparib: Eligible participants who initiated treatment with talazoparib for HER2- mBC gBRCA 1/2m on or after 01-Jan-2018 were included.
Arm/Group | Talazoparib
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.64 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3
  White | 18
  Other | 11
  Unknown/Undocumented | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Unknown | 31
Number of Participants According to Subtypes of Breast Cancer [Count of Participants; unit: Participants] — Number of participants with HER2- mBC gBRCA 1/2m were classified according to their sub-types as HR+/HER2- and triple negative breast cancer (TNBC) were reported.
  Participants
    HR+/HER2 - | 26
    TNBC | 7
Number of Participants According to gBRCA Mutation Type [Count of Participants; unit: Participants] — Number of participants classified according to gBRCA mutation as breast cancer susceptibility gene 1(BRCA 1), breast cancer susceptibility gene 2 (BRCA 2), breast cancer susceptibility not otherwise specified (BRCA mutation NOS) were reported.
  Participants
    BRCA 1 mutation identified | 11
    BRCA 2 mutation identified | 21
    BRCA mutation NOS | 1
Line of mBC Therapy in Which Talazoparib was Administered [Count of Participants; unit: Participants] — Number of participants were classified according to line of mBC therapy in which talazoparib was initiated were reported.
  Participants
    First | 5
    Second | 6
    Third | 9
    Fourth | 3
    Fifth | 2
    Sixth | 3
    Seventh | 2
    Eighth | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (TTF) for Talazoparib
Description: TTF was defined as the time from initiation of talazoparib to discontinuation for any reason, which included disease progression, treatment toxicity, and death. Participants who were still on therapy at the end of follow-up (earliest of last participant-level structured or abstracted activity [i.e., the last record of participant vitals, medication administrations, or reported laboratory tests/results, or abstracted end date of oral medications] or date of data cut-off [30 September 2020]) were censored. Index date was defined as the date first talazoparib-containing line of therapy between 01-Jan-2018 to 30-Sep-2020. Median was analyzed using the Kaplan-Meier method.
Time Frame: Index date up to talazoparib discontinuation or at the end of follow-up or date of data cut-off (30-September-2020), maximum up to approximately 2.9 years; data retrieved and studied approximately 6.14 months of this study
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 33
Months | 5.5 [2.1 to 10.5]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study
Description: Minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Arm/Group | Talazoparib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT05141708/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT05141708/SAP_001.pdf